CLINICAL TRIAL: NCT04988256
Title: A Randomized Controlled Pilot Trial of Cyclosporine Vs Steroids in DRESS
Brief Title: Cyclosporine Vs Steroids in DRESS
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Scott Worswick, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-20-00118
Record Dates: First submitted 2021-06-24; First posted 2021-08-03 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-12

CONDITIONS: DRESS Syndrome; Drug-Induced Hypersensitivity Syndrome
MeSH Terms: conditions — Drug Hypersensitivity Syndrome | interventions — Cyclosporine; Methylprednisolone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyclosporine (Active Comparator): All Patients start with 5 mg/kg/day (3 mg/kg/day if renal impairment) PO divided bid for 7 days (or IV if patient is NPO)
  1. If complete resolution, stop cyclosporine and monitor closely for relapse
     a. If patient relapses, give 5 (3 if renal impairment) mg/kg/day PO divided bid PO for 7 days
     i. If down-trending, start oral taper regimen
     ii. If not down-trending, switch to steroid arm
  2. If >25% improvement and labs are down-trending, start the oral taper regimen.
  3. If 0-25% improvement, give 5 (3 if renal impairment) mg/kg/day PO divided bid for 3 days
     1. If down-trending, start oral taper regimen
     2. If not down-trending, switch to steroid arm
  4. If no improvement or up-trending labs at 7 days, switch to steroid arm
  Oral Taper Regimen set as 3 mg/kg PO divided bid for 14 days, then 2 mg/kg PO divided bid for 20 days. If renal impairment, oral taper regimen set as 2 mg/kg PO divided bid for 14 days, then 1 mg/kg PO divided bid for 20 days
  Interventions: Drug: Cyclosporine
- Corticosteroids (Experimental): All Patients start with 500 mg IV Methylprednisolone for 3 days
  1. If >25% improvement (must be >25% in all involved organs), start the taper regimen 2. If 0-25% improvement (in ≥1 involved internal organ), give 500 mg IV Methylprednisolone for 4 days
  1. If no improvement, switch to cyclosporine arm of treatment
  2. If 0-25% improvement, give 500 mg IV Methylprednisolone for 3 days
  i. If labs are down-trending, start the taper regimen
  ii. If labs are not down-trending, switch to cyclosporine arm of the study
  c. If >25% improvement, start the taper regimen
  Taper Regimen set as:
  1. 125 mg IV Methylprednisolone x3 days
  2. 1.2 mg/kg PO prednisone x1 week
  3. 1 mg/kg PO prednisone x1 week
  4. 0.8 mg/kg PO prednisone x1 week
  5. 0.6 mg/kg PO prednisone x1 week
  6. 0.4 mg/kg PO prednisone x1 week
  7. 0.2 mg/kg PO prednisone x1 week
  8. 0.1 mg/kg PO prednisone x1 week
  9. 0.05 mg/kg PO prednisone x1 week
  Interventions: Drug: Methylprednisolone and Prednisone

INTERVENTIONS:
Drug: Cyclosporine — Patients randomized to cyclosporine will be treated as mentioned under "Arm/Group Description"
  Arms: Cyclosporine
Drug: Methylprednisolone and Prednisone — All patients randomized to steroids will initially be treated with IV methylprednisolone and eventually started on an oral prednisone taper.
  Arms: Corticosteroids

SUMMARY:
Current treatments for patients with drug reaction with eosinophilia and systemic symptoms (DRESS) include supportive care, steroids and cyclosporine. No randomized controlled trial (RCT) exists in comparing these treatments and all available literature comes in the form of case reports and case series. These two treatments are considered standard of care and this trial seeks only to compare outcomes of DRESS between these two therapies. No additional labs, therapies or procedures will be used apart from those that are routinely done for patients with this diagnosis.

This will be a pilot study to determine efficacy of the two therapies with particular endpoints in mind so that the investigators can study the safety of these two therapies in patients with DRESS.

Data suggests a potential benefit for adults with DRESS using either steroids or cyclosporine but the investigators are seeking a comparison of efficacy of these two therapies. The study population will include adults with a Registry of Severe Cutaneous Adverse Reaction (RegiSCAR) score of greater than 4 (i.e. a likely diagnosis of DRESS). The investigators will exclude patients with sepsis, active Hepatitis B or C, active tuberculosis, a documented allergy to steroids or cyclosporine, and patients with an estimated glomerular filtration rate (eGFR) < 30 (unless on dialysis in which case the participants will be included).

DETAILED DESCRIPTION:
Current treatments for patients with drug reaction with eosinophilia and systemic symptoms (DRESS) include supportive care, steroids, cyclosporine and to a lesser extent, intravenous immunoglobulin (IVIG). Regarding IVIG, a recent case series suggests no improved benefit in adults. No randomized controlled trial (RCT) exists in comparing these treatments and all available literature comes in the form of case reports and case series. These two treatments are considered standard of care and this trial seeks only to compare outcomes of DRESS between these two therapies. No additional labs, therapies or procedures will be used apart from those that are routinely done for patients with this diagnosis.

This will be a pilot study to determine efficacy of the two therapies with particular endpoints in mind so that the investigators can study the safety of these two therapies in patients with DRESS. Hopefully, this study will allow the investigators to better power a full prospective trial in the future.

This is a potentially life-threatening severe cutaneous adverse reaction (SCAR) with significant potential morbidity. Data suggests a potential benefit for adults with DRESS using either steroids or cyclosporine but the investigators are seeking a comparison of efficacy of these two therapies. The study population will include adults with a Registry of Severe Cutaneous Adverse Reaction (RegiSCAR) score of greater than 4 (i.e. a likely diagnosis of DRESS). The investigators will exclude patients with sepsis, active Hepatitis B or C, active tuberculosis, a documented allergy to steroids or cyclosporine, and patients with an estimated glomerular filtration rate (eGFR) < 30 (unless on dialysis in which case the participants will be included).

Participants will be randomized using a randomization protocol at all sites. Primary endpoints will include percentage of participants with complete or near complete resolution of organ involvement as well as erythema resolution at day 7 and day 30.

Secondary endpoints will be:

1. fever presence, resolution of facial edema, resolution of pruritus, lymphadenopathy, eosinophil count at days 7 and 30
2. days of hospitalization
3. mortality at days 7, 30 and 90
4. viral reactivation at days 30, 60 and 90
5. those with autoimmune development by day 30 and day 90
6. 30 day re-admission rate.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a RegiSCAR score of greater than 4 (i.e a likely diagnosis of DRESS)

Exclusion Criteria:

* Active sepsis
* Active hepatitis B or C
* Active tuberculosis
* Documented allergy to steroids or cyclosporine
* Estimated glomerular filtration rate (eGFR) < 30 (unless on dialysis, in which case they will be included)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with complete or near complete resolution of organ involvement at day 30, on steroid therapy and cyclosporine therapy | Day 7
  Measured by the following quantitative metrics:
  * Creatinine within 1.25x of baseline or upper limit of normal, whichever is higher
  * Aspartate Aminotransferase (AST) within 1.5x of baseline or upper limit of normal, whichever is higher
  * Troponin-T, Creatine Kinase Myocardial Band (CK-MB), Pro B-type Natriuretic Peptide (Pro-BNP), and lipase within 1.25x of baseline or upper limit of normal, whichever is higher
  * Resolution of interstitial pneumonitis on chest x-ray
Percentage of patients with complete or near complete resolution of organ involvement at day 30, on steroid therapy and cyclosporine therapy | Day 30
  Measured by the following quantitative metrics:
  * Creatinine within 1.25x of baseline or upper limit of normal, whichever is higher
  * Aspartate Aminotransferase (AST) within 1.5x of baseline or upper limit of normal, whichever is higher
  * Troponin-T, Creatine Kinase Myocardial Band (CK-MB), Pro B-type Natriuretic Peptide (Pro-BNP), and lipase within 1.25x of baseline or upper limit of normal, whichever is higher
  * Resolution of interstitial pneumonitis on chest x-ray
Percentage of patients with complete or near complete resolution of erythema at day 7, on steroid therapy and cyclosporine therapy | Day 7
  Clinical measurement of erythema
Percentage of patients with complete or near complete resolution of erythema at day 30, on steroid therapy and cyclosporine therapy | Day 30
  Clinical measurement of erythema

SECONDARY OUTCOMES:
Percentage of patients with resolution of fever | Day 7
  Less than 38 degrees Celsius for at least 24 hours
Percentage of patients with resolution of fever | Day 30
  Less than 38 degrees Celsius for at least 24 hours
Percentage of patients with resolution of facial edema | Day 7
  Clinical resolution of edema for at least 24 hours
Percentage of patients with resolution of facial edema | Day 30
  Clinical resolution of edema for at least 24 hours
Percentage of patients with resolution of pruritus | Day 7
  Resolution for at least 24 hours
Percentage of patients with resolution of pruritus | Day 30
  Resolution for at least 24 hours
Percentage of patients with resolution of lymphadenopathy | Day 7
  Clinical resolution of lymphadenopathy for at least 24 hours
Percentage of patients with resolution of lymphadenopathy | Day 30
  Clinical resolution of lymphadenopathy for at least 24 hours
Absolute eosinophil proportion compared to peak value | Day 7
  Proportion of absolute eosinophils
Absolute eosinophil proportion compared to peak value | Day 30
  Proportion of absolute eosinophils
Patients with autoimmune disease development | Day 30
  Measured by titers of autoimmune markers (Antinuclear Antibody (ANA), Thyroid Stimulating Hormone (TSH)) compared to baseline
Patients with autoimmune disease development | Day 90
  Measured by titers of autoimmune markers (Antinuclear Antibody (ANA), Thyroid Stimulating Hormone (TSH)) compared to baseline
Total days of hospitalization after initial dermatology consult | 0-120 days
  Number of days
Viral reactivation | Day 30
  Measured by titers of Human Herpesvirus 6 (HHV6), Cytomegalovirus (CMV), and Epstein-Barr Virus (EBV)
Viral reactivation | Day 60
  Measured by titers of Human Herpesvirus 6 (HHV6), Cytomegalovirus (CMV), and Epstein-Barr Virus (EBV)
Viral reactivation | Day 90
  Measured by titers of Human Herpesvirus 6 (HHV6), Cytomegalovirus (CMV), and Epstein-Barr Virus (EBV)
Mortality | Day 7
  Proportion of patient mortality
Mortality | Day 30
  Proportion of patient mortality
Mortality | Day 90
  Proportion of patient mortality
30-day readmission rate | Day 30
  Proportion of patients re-admitted to the hospital within 30 days of discharge

CONTACTS AND LOCATIONS:
Locations (1):
- USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No